CLINICAL TRIAL: NCT02623335
Title: Navigating High Risk Surgery: Empowering Older Adults to Ask Questions That Inform Decisions About Surgical Treatment
Brief Title: PCORI-1502-27462 Navigating High Risk Surgery: Empowering Older Adults to Ask Questions That Inform Decisions About Surgical Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of California, San Francisco (Other); Brigham and Women's Hospital (Other); New Jersey Medical School (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2015-1375
Record Dates: First submitted 2015-11-24; First posted 2015-12-07 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Communication
Keywords: patient decision making; surgical decision making; question prompt list; shared decision making; decision support techniques
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QPL (question prompt list) brochure (Experimental): Patients were mailed the QPL (question prompt list) prior to their appointment with an enrolled surgeon.
  Interventions: Other: QPL (question prompt list) brochure
- Usual care (No Intervention): The investigators observed that usual care included informed consent and a surgeon-directed deliberative phase in which surgeons presented their own evaluation of the trade-offs and goals of the proposed intervention.

INTERVENTIONS:
Other: QPL (question prompt list) brochure — The QPL intervention includes the QPL intervention brochure, plus a letter from the surgeon encouraging its use during the upcoming office visit. Intervention materials will be mailed in advance of the patient's appointment with an enrolled surgeon.
  Arms: QPL (question prompt list) brochure

SUMMARY:
The investigators will perform a multi-site cluster randomized trial that uses a stepped-wedged design to compare the effectiveness of a Question Prompt List (QPL) intervention to usual care for patients considering high-risk vascular (peripheral, cardiac, neuro) and oncologic operations. This 24-month study will use a time-dependent cluster randomization plan within each of the five study sites: the investigators will randomly assign time points for surgeons who perform high risk operations to cross over from usual care to QPL intervention. Study staff will audiotape the conversation between the patient and surgeon during one preoperative clinic visit; administer surveys to patients and family members at 24 hours, 6 weeks and 12 weeks after that visit; and record surgical decisions, treatments received and associated outcomes. The investigators will use stratified purposeful sampling to identify a subset of patients in each study arm who have experienced serious complications for qualitative interviews.

DETAILED DESCRIPTION:
To answer the research question, "Could a patient-driven approach that improves decision making and informs postoperative expectations have more effectiveness than the current surgeon-directed preoperative conversation?" the investigators will conduct a multi-site randomized controlled trial of the question prompt list intervention (QPL) for high risk surgery that will:

1. Compare the effectiveness of the intervention relative to usual care on the extent of patient engagement in decision-making for high risk surgery. (Aim 1)
2. Compare the effectiveness of the intervention relative to usual care on treatment choice and on psychological well-being and post-treatment regret for patients and family members. (Aim 2)
3. Compare the effectiveness of the intervention relative to usual care on interpersonal and intrapersonal conflict relating to treatment decisions and subsequent treatments received. (Aim 3)

The overall goals of the study are to help patients and families:

1. make treatment decisions aligned with their values and goals;
2. anticipate and make sense of postoperative outcomes; and
3. experience less postoperative conflict about treatment of serious complications.

Enrolled surgeons will be grouped based on self-report of their clinic practices. "Visit 1 Surgeons" typically have a treatment decision making conversation with patients at their initial new patient consult. For enrolled patients of these surgeons, we will audio-record their first consult visit. "Visit 2 Surgeons" typically do not have treatment decision making discussions at the initial visit- this discussion is generally delayed until a follow up appointment, after additional testing or review of medical records. The return/second visit of enrolled patients under the care of Visit 2 Surgeons will be recorded.

When a surgeon is in the usual care arm, patients will receive the current standard for surgical decision-making. Once an enrolled surgeon has crossed into the intervention arm, the research team will mail the QPL intervention to all of the surgeon's new consult patients (for Visit 1 Surgeons) or returning/2nd consult patients (for Visit 2 Surgeons) about a week prior to their scheduled consultation, regardless of study eligibility. The QPL intervention includes the QPL intervention brochure, plus a letter from the surgeon encouraging its use during the upcoming office visit. Eligible patients will be identified by clinic staff and interested patients will be approached once they arrive in clinic (they will not receive information about the study prior to their clinic appointment because this information could interfere with the QPL intervention).

Patients in the usual care arm will receive the current standard for surgical decision-making. The investigators have observed that usual care includes informed consent and a surgeon-directed deliberative phase in which surgeons present their own evaluation of the trade-offs and goals of the proposed intervention. Although this deliberation occurs in front of patients and families, assumptions about the value of specific outcomes are surgeon-generated and not specifically linked to patient preferences. For these reasons, the investigators believe comparing the intervention to usual care is suitable. In addition, question prompt lists are currently available online and are not distributed by the surgeon. Patients can obtain and use the lists if they so choose on their own (although most do not). Additionally, question prompt lists have been shown to be safe and effective in previous studies in similar but not identical clinical situations.

Surgeons will be randomly assigned within each site to change from usual care to the QPL intervention at different study wave time points. Prior to study start the investigators will conduct step-wise randomization using a computer-generated randomization schedule to determine the crossover wave timing among surgeons. Surgeon cross-over from usual care to intervention will occur in one direction only and each within-site change will occur once every four months. Surgical clinics will be contacted one month prior to intervention implementation to confirm and execute implementation processes and to start mailing the QPL intervention to patients with office visits scheduled on or after the first day of intervention transition. A 2-week hiatus in data collection at the start of the cross over will be instituted in the transition clinics to ensure patients in the intervention group have had the opportunity to receive the intervention mailing. Surgeons who have crossed over to the intervention group will be notified when the QPL intervention has been implemented in their clinic and will be encouraged with bi-weekly email or text reminders to support patient use of the question list during clinical encounters with patients discussing surgical treatment options.

For patients in both the usual care and intervention arms: Surgeons who perform high risk operations and have agreed to participate will help to identify new or returning patients (depending on their previously reported practice pattern) coming to an outpatient visit to discuss a major surgical procedure. If a patient consents to the study, study staff will audio record one conversation (T0) between the attending surgeon and patient and accompanying family member. Study staff will meet with the patient prior to starting the audio recording to obtain consent. If there is a family member present at the appointment and he or she would like to participate in study activities, study staff will obtain consent from them as well. If a resident/surgical trainee or additional family members and caretakers are present, study staff will obtain verbal permission to audio record the resident and all others present. Study staff will wait until the surgeon enters the room and then turn on the digital audio recorder. Once the audio recorder has been turned on, the research team member will leave the room and return once the meeting between the patient and surgeon is complete to terminate and collect the audio recording.

Study staff will conduct follow-up phone calls to administer surveys to the patient and family member (if they have enrolled) within 12-72 hours of the patient's audio-recorded treatment decision-making visit (T1). After the visit with the surgeon, the patient's treatment plan will be determined by chart review and confirmed with the surgeon or clinic nurse. Administration of the second and third surveys (T2 and T3) will be linked to the patient's treatment plan. For patients who are scheduled for surgery, surveys will be administered via telephone to the patient and family member 1-2 (T2) weeks after surgery and 6-8 (T3) weeks after surgery. Based on previous study in this patient population and clinical setting, the median time between the patient's preoperative visit with the surgeon and surgery is 31 days. If the patient is unable to participate in study activities, enrolled family members will still be asked to complete study activities. Patients who did not have a family member enroll along with them and who are unable to participate in study activities post-operatively will be considered lost to follow up. For patients who have non-operative treatment; e.g., medical treatment (chemotherapy, pulmonary rehab) or observation (active surveillance, no surgical procedure scheduled), study staff will administer surveys between 6 and 8 weeks (T2) and again between 12 and 14 (T3) weeks after the patient's audio-recorded treatment decision-making visit with the surgeon. This will roughly approximate the time frame for study activities for patients who have surgery. Patients and family members will also be allowed to complete follow up surveys (T2 and T3) by web survey or mail, if they prefer, though phone surveys will likely be the primary data collection method, based on prior research.

Some patients of Visit 1 Surgeons will need additional testing (CT scan, PET scan, stress test) before a treatment decision can be made. These patients and their family members will complete the initial study activities (audio recording of the initial visit with a surgeon (T0) and survey at 12-72 hours (T1)). Study staff will not audio record a second (return) visit with the surgeon or repeat the post visit survey (T1). The second and third surveys will be linked to the treatment decision after this second interaction with the surgeon: T2: 1-2 weeks postoperatively and T3: 6-8 weeks postoperatively, or T2: 6-8 and T3:12-14 weeks after the second interaction with the surgeon for those who have non-operative treatment. In some cases surgeons will telephone the patient after additional testing to develop a treatment plan. Study staff will not audio record this interaction. Study staff will use careful chart review and communication with the surgeon and/or his/her clinical staff for these patients to accurately target the timing of subsequent study activities. After the final survey is completed study staff will use chart abstraction to identify and record treatments received and postoperative complications.

Study staff will use chart review immediately after the patient meets with the surgeon (T0) and again after the final survey (T3) has been completed to record clinical data, treatments received and outcomes of treatment. Study staff will also screen charts of enrolled patients weekly in order to confirm treatment plan which may be unclear at the time of their audio-recorded treatment decision-making visit and is critically important to timing of subsequent data collection. Data collected will be limited to clinical information pertaining to surgical care from audio-recorded treatment decision-making visit through to administration of the final survey (T3).

To investigate Aim 3, the investigators will use a qualitative study design to compare interpersonal and intrapersonal conflict between study arms as it relates to the phenomenon of surgical buy in-when the surgeon believes that the patient has agreed to the operative procedure as well as all possible postoperative care. Conflict between surgeons and patients and/or family members about additional invasive procedures occurs in the uncommon setting of serious postoperative complications but may be affected by the QPL intervention, which includes questions about "What happens if things go wrong?" and specific question prompts about advance directives. Thus, investigators will use stratified purposeful sampling to identify a subset of patients who have experienced serious postoperative complications in each study arm, as determined by chart review. Serious complications include prolonged hospitalization (more than 8 days postoperatively), prolonged length of stay in intensive care (greater than 3 days), prolonged mechanical ventilation, myocardial infarction, major cerebrovascular accident, new onset dialysis or death. Study staff will use chart review at T3 (12-14 weeks, roughly 6 weeks after surgery) to identify patients who have had serious complications and ask them and/or their family members to participate in a face-to-face qualitative interview. The investigators are planning for 3-7 interviews at each study site and anticipate no more than 10 at each site. Not all patients who consent to Aims 1 and 2 of the study will participate in Aim 3.

For patients and family members who agree to be interviewed, a trained Qualitative Interviewer will conduct the interview. The interviewer will meet the patient and family member at a convenient and private location of their choosing for an in-person interview. Patients and family members will have the choice to conduct the interview jointly or separately. Study investigators have employed this technique in previous studies and successfully interviewed study participants and family members in their homes or at the medical center in a private room at the time of a follow up medical appointment. Interviews will generally not be conducted over the telephone as this limits the ability of the interviewer to respond to non-verbal cues. Interviews will last up to one hour.

ELIGIBILITY:
Surgeons

Inclusion Criteria:

* Consenting surgeons at participating hospital sites who practice vascular, cardiothoracic, hepatobiliary, colorectal, urologic, gynecologic, head and neck or neurosurgery
* Regularly see patients preoperatively in the surgical clinic
* Perform high risk operations on older patients with multiple comorbid conditions

Exclusion Criteria:

* Exclusively perform minimally invasive surgery (laparoscopy), endocrine or breast surgery as these procedures are not typically considered "high risk"
* Patient panel is not generally comprised of older adults considering high risk procedures

Patients

Inclusion Criteria:

* Age 60 and older
* One or more chronic conditions from a list comprised of those included in the Charlson Comorbidity Index with 9 additional conditions included due to their saliency to surgical decision making
* Have an upcoming outpatient consultation with an enrolled surgeon to discuss treatment for a vascular or oncologic problem that can be treated with a high risk operation
* English speaking and Spanish-speaking patients who require an interpreter will be included

Exclusion Criteria:

* Lack decision-making capacity
* Deemed too physically or mentally ill to participate by their surgeon or clinic nurse
* Self-report that their vision or literacy skills are too poor to read a newspaper
* Cannot speak either English or Spanish with the fluency required to have a valid medical decision-making conversation as the QPL is currently only available in English and Spanish (Spanish speaking patients who require an interpreter to speak with their surgeon will be included)
* Participating surgeons may also choose to exclude specific patients for study participation based on their own concerns about the patient participating in the study, for example patients who have urgent surgical needs or don't actually have a surgical problem

Family members

Inclusion Criteria:

* Family member (patient participant) is enrolled in the study
* Present at time of patient enrollment in study

Exclusion Criteria:

* Lack decision-making capacity
* Self-report that their vision or literacy skills are too poor to read a newspaper
* Cannot speak either English or Spanish with the fluency required to have a valid medical decision-making conversation as the QPL is currently only available in English and Spanish (Spanish speaking patients who require an interpreter to speak with the surgeon will be included)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2016-02; Primary Completion 2018-11-15 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Schwarze, MD, MPP, FACS, Principal Investigator — University of Wisconsin, Madison; Emily Finlayson, MD, MS, Principal Investigator — University of California, San Francisco; Zara Cooper, MD, MSc, Principal Investigator — Brigham and Women's Hospital; Anne Mosenthal, MD, Principal Investigator — Rutgers University; Ana Berlin, MD, MPH, Principal Investigator — Rutgers University; Karen Brasel, MD, MPP, Principal Investigator — Oregon Health and Science University

REFERENCES:
- [Derived] Stalter LN, Baggett ND, Hanlon BM, Buffington A, Kalbfell EL, Zelenski AB, Arnold RM, Clapp JT, Schwarze ML. Identifying Patterns in Preoperative Communication about High-Risk Surgical Intervention: A Secondary Analysis of a Randomized Clinical Trial. Med Decis Making. 2023 May;43(4):487-497. doi: 10.1177/0272989X231164142. Epub 2023 Apr 10. PMID 37036062
- [Derived] Baggett ND, Schulz K, Buffington A, Marka N, Hanlon BM, Zimmermann C, Tucholka J, Fox D, Clapp JT, Arnold RM, Schwarze ML. Surgeon Use of Shared Decision-making for Older Adults Considering Major Surgery: A Secondary Analysis of a Randomized Clinical Trial. JAMA Surg. 2022 May 1;157(5):406-413. doi: 10.1001/jamasurg.2022.0290. PMID 35319737
- [Derived] Kalbfell E, Kata A, Buffington AS, Marka N, Brasel KJ, Mosenthal AC, Cooper Z, Finlayson E, Schwarze ML. Frequency of Preoperative Advance Care Planning for Older Adults Undergoing High-risk Surgery: A Secondary Analysis of a Randomized Clinical Trial. JAMA Surg. 2021 Jul 1;156(7):e211521. doi: 10.1001/jamasurg.2021.1521. Epub 2021 Jul 14. PMID 33978693
- [Derived] Schwarze ML, Buffington A, Tucholka JL, Hanlon B, Rathouz PJ, Marka N, Taylor LJ, Zimmermann CJ, Kata A, Baggett ND, Fox DA, Schmick AE, Berlin A, Glass NE, Mosenthal AC, Finlayson E, Cooper Z, Brasel KJ. Effectiveness of a Question Prompt List Intervention for Older Patients Considering Major Surgery: A Multisite Randomized Clinical Trial. JAMA Surg. 2020 Jan 1;155(1):6-13. doi: 10.1001/jamasurg.2019.3778. PMID 31664452
- [Derived] Taylor LJ, Rathouz PJ, Berlin A, Brasel KJ, Mosenthal AC, Finlayson E, Cooper Z, Steffens NM, Jacobson N, Buffington A, Tucholka JL, Zhao Q, Schwarze ML. Navigating high-risk surgery: protocol for a multisite, stepped wedge, cluster-randomised trial of a question prompt list intervention to empower older adults to ask questions that inform treatment decisions. BMJ Open. 2017 May 29;7(5):e014002. doi: 10.1136/bmjopen-2016-014002. PMID 28554911

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Surgeons at 5 sites were recruited by email and in-person contact. After they were consented, their patients were screened for eligibility and approached in clinic to discuss study participation.
Groups:
- QPL (Question Prompt List) Brochure: Patients were mailed the QPL (question prompt list) prior to their appointment with an enrolled surgeon.
  QPL (question prompt list) brochure: The QPL intervention included the QPL intervention brochure, plus a letter from the surgeon encouraging its use during the upcoming office visit. Intervention materials were mailed in advance of the patient's appointment with an enrolled surgeon.
Period: Overall Study
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care
Started | 223 | 223
T0 Audio Recording (Day of Consultation) | 223 | 222
T1 Survey (24-48 Hours) | 216 | 214
T2 Survey (6-8 Weeks) | 199 | 192
T3 Survey (12-14 Weeks) | 196 | 187
Completed | 196 | 187
Not Completed | 27 | 36
Not completed — Death | 8 | 7
Not completed — Lost to Follow-up | 15 | 23
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care | Total
Number analyzed (Participants) | 223 | 223 | 446
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 24 | 65
  >=65 years | 182 | 199 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.01 (6.67) | 72.59 (7.34) | 71.8 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 93 | 197
  Male | 119 | 130 | 249
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 13 | 31
  Not Hispanic or Latino | 197 | 197 | 394
  Unknown or Not Reported | 8 | 13 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 11 | 4 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 18 | 18 | 36
  White | 178 | 182 | 360
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 223 | 223 | 446

OUTCOME MEASURES:

1. Primary Outcome: Patient Engagement in Decision Making Measured by Clinic Visit Transcript Coding for Number of and Types of Questions Raised
Description: Patient engagement in decision making was measured by coding the transcript for the patient's clinic visit, using a pre-defined coding scheme that focused on the number and types of questions raised in the audio-recorded treatment decision-making visit. The types of questions that were coded were options questions, expectations questions, risks questions and advance directive questions.
Time Frame: Within 2 hours of enrollment in the study
Population: Due to instances when a full audio recording of the clinic visit was not available, the number of participants analyzed differs from the number of total arm participants.
Measure: Count of Participants; unit: Participants
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care
Number analyzed (Participants) | 216 | 219
Participants
  Options question asked (2 or more) | 68 | 55
  Expectations question asked (2 or more) | 95 | 89
  Risks question asked (2 or more) | 35 | 36
  Advance Directives question asked (1 or more) | 3 | 0
Statistical Analysis 1: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; Options questions; Test type: Superiority; p = 0.353, Mixed Models Analysis; Odds Ratio (OR) = 1.32
Statistical Analysis 2: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; Expectations questions; Test type: Superiority; p = 0.923, Mixed Models Analysis; Odds Ratio (OR) = 0.97
Statistical Analysis 3: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; Risks questions; Test type: Superiority; p = 0.255, Mixed Models Analysis; Odds Ratio (OR) = 1.41
Statistical Analysis 4: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; Advance directives questions; Test type: Superiority; p = 0.094, Mixed Models Analysis; Odds Ratio (OR) = 239047259

2. Primary Outcome: Change in Illness-related Stress Measured by Participant Self-report on MYCaW Instrument
Description: Changes in concerns and well-being were measured using the self-report instrument Measure Yourself Concerns and Well-being (MYCaW) instrument. The minimum value for differences in this scale is -6 and maximum value is 6. Higher scores indicate that problems and concerns have diminished.
Time Frame: 24-48 hours after enrollment, 6-8 weeks post-enrollment and 3-4 months post-enrollment
Population: The number of participants analyzed differs from the number of total arm participants due to a low rate of survey or item non-response.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care
Number analyzed (Participants) | 136 | 154
change in score on a scale
  Change in scores between T2 and T1: number analyzed (Participants) | 117 | 123
  Change in scores between T2 and T1 | -1.49 (2.76) | -1.6 (2.41)
  Change in scores between T3 and T1: number analyzed (Participants) | 110 | 124
  Change in scores between T3 and T1 | -1.88 (2.66) | -1.73 (2.49)
Statistical Analysis 1: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; Change in scores between T2 and T1; Test type: Superiority; p = 0.84, Mixed Models Analysis; Effect estimate = -0.04
Statistical Analysis 2: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; Change in scores between T3 and T1; Test type: Superiority; p = 0.645, Mixed Models Analysis; Effect estimate = -0.15

3. Primary Outcome: Perceived Self-efficacy in Patient-physician Interactions Measured by Participant Self-report on the PEPPI-5 Scale
Description: Perceived self-efficacy in patient-physician interactions was measured by participant self-report, using the 5-item Perceived Efficacy in Patient-Physician Interactions (PEPPI-5) scale. Maximum value for this scale is 25 and minimum is 0. Higher scores indicate greater self-efficacy.
Time Frame: 24-48 hours after enrollment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care
Number analyzed (Participants) | 208 | 202
score on a scale | 21.64 (3.38) | 21.45 (3.31)
Statistical Analysis 1: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; Test type: Superiority; p = 0.411, Mixed Models Analysis; Effect estimate = -0.37

4. Primary Outcome: Post-treatment Regret Measured by a Specific Participant Self-report Survey Item
Description: Post-treatment regret was assessed by the following participant self-report survey item: "Looking back, is there anything about your treatment that you would do differently?"
Time Frame: 3-4 months post-enrollment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care
Number analyzed (Participants) | 205 | 209
Participants
  Had regret | 61 | 48
  No regret | 144 | 161
Statistical Analysis 1: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; Test type: Superiority; p = 0.412, Mixed Models Analysis; Odds Ratio (OR) = 1.39

5. Secondary Outcome: Participant Autonomy Support Measured by Self-report on the HCCQ Instrument
Description: Participant autonomy support was assessed using the self-report measure Health Care Climate Questionnaire (HCCQ). The minimum value for this scale is 1 and the maximum value is 7. Higher scores indicate greater perceived autonomy support.
Time Frame: 24-48 hours after enrollment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care
Number analyzed (Participants) | 208 | 202
score on a scale | 6.39 (0.8) | 6.5 (0.65)
Statistical Analysis 1: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; Test type: Superiority; p = 0.009, Mixed Models Analysis; Effect estimate = -0.25

6. Secondary Outcome: Patient and Family Psychological Well-being Measured by Self-report on the PROMIS Psychosocial Illness Impact- Positive Scale
Description: Changes in family psychological well-being were assessed by participant self-report using the Patient Reported Outcomes Measurement Information System (PROMIS) Psychosocial Illness Impact- Positive scale. The minimum value for this scale is 4 and the maximum is 16. Higher values indicate better well-being.
Time Frame: 6-8 weeks post-enrollment, 3-4 months post-enrollment post-enrollment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care
Number analyzed (Participants) | 179 | 175
score on a scale
  6-8 weeks post-enrollment (T2): number analyzed (Participants) | 179 | 168
  6-8 weeks post-enrollment (T2) | 12.92 (3.12) | 13.52 (3.03)
  3-4 months post-enrollment post-enrollment (T3): number analyzed (Participants) | 176 | 175
  3-4 months post-enrollment post-enrollment (T3) | 12.95 (3.05) | 13.64 (2.6)
Statistical Analysis 1: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; 6-8 weeks post-enrollment (T2); Test type: Superiority; p = 0.106, Mixed Models Analysis; Effect estimate = -0.72
Statistical Analysis 2: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; 3-4 months post-enrollment post-enrollment (T3); Test type: Superiority; p = 0.007, Mixed Models Analysis; Effect estimate = -1.12

7. Secondary Outcome: Patient and Family Psychological Well-being Measured by Self-report on the PROMIS Psychosocial Illness Impact- Negative Scale
Description: Changes in family psychological well-being were assessed by participant self-report using the Patient Reported Outcomes Measurement Information System (PROMIS) Psychosocial Illness Impact- Negative scale. Minimum value for this scale is 4 and maximum is 20. Higher values indicate worse well-being.
Time Frame: 6-8 weeks post-enrollment, 3-4 months post-enrollment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care
Number analyzed (Participants) | 179 | 176
score on a scale
  6-8 weeks post-enrollment (T2): number analyzed (Participants) | 165 | 167
  6-8 weeks post-enrollment (T2) | 6.92 (3.45) | 6.47 (2.83)
  3-4 months post-enrollment (T3) | 7.05 (3.67) | 6.25 (2.77)
Statistical Analysis 1: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; 6-8 weeks post-enrollment (T2); Test type: Superiority; p = 0.034, Mixed Models Analysis; Effect estimate = 0.97
Statistical Analysis 2: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; 3-4 months post-enrollment (T3); Test type: Superiority; p = 0.019, Mixed Models Analysis; Effect estimate = 1.12

8. Secondary Outcome: Patient and Family Psychological Well-being Measured by Self-report on the PROMIS Anxiety 4a Scale
Description: Changes in family psychological well-being were assessed by participant self-report using the Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety 4a scale. Minimum value for this scale is 4 and maximum is 20. Higher values indicate worse well-being.
Time Frame: 6-8 weeks post-enrollment, 3-4 months post-enrollment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care
Number analyzed (Participants) | 180 | 180
score on a scale
  6-8 weeks post-enrollment (T2): number analyzed (Participants) | 169 | 166
  6-8 weeks post-enrollment (T2) | 7.57 (3.57) | 7.18 (3.43)
  3-4 months post-enrollment post-enrollment (T3) | 7.18 (3.5) | 6.76 (3.26)
Statistical Analysis 1: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; 6-8 weeks post-enrollment (T2); Test type: Superiority; p = 0.022, Mixed Models Analysis; Effect estimate = 1.16
Statistical Analysis 2: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; 3-4 months post-enrollment post-enrollment (T3); Test type: Superiority; p = 0.053, Mixed Models Analysis; Effect estimate = 0.94

9. Secondary Outcome: Number of Participants Who Had Surgery During the Study Period
Description: The total number of participants who had surgery during the study period was tracked through a patient chart review.
Time Frame: From enrollment to end of data collection 3-4 months later
Population: The number of participants analyzed differs from the number of total arm participants due to a low rate of participant drop out from the chart review study activity.
Measure: Count of Participants; unit: Participants
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care
Number analyzed (Participants) | 220 | 220
Participants | 135 | 139

10. Secondary Outcome: Physician Engagement With Patient Measured by Clinic Visit Transcript Coding Using OPTION Coding System
Description: Physician engagement with patient was measured by coding the transcript for the patient's clinic visit, using the Observing Patient Involvement in Decision Making instrument (OPTION) scale. Minimum value for this scale is 0 and maximum is 100. Higher scores indicate increased shared decision making.
Time Frame: Within 2 hours of enrollment in the study
Population: The number of participants analyzed differs from the number of total arm participants due to a low number of cases where full audio recording of clinic visit was unavailable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care
Number analyzed (Participants) | 216 | 219
score on a scale | 34.26 (21.56) | 31.03 (19.84)
Statistical Analysis 1: Comparison: QPL (Question Prompt List) Brochure vs Usual Care; Test type: Superiority; p = 0.07, Mixed Models Analysis; Effect estimate = 5.04

ADVERSE EVENTS:
Time Frame: Up to approximately 6 months following enrollment
Arm/Group | QPL (Question Prompt List) Brochure | Usual Care
All-Cause Mortality (participants affected / at risk) | 8/223 | 7/223
Serious Adverse Events (participants affected / at risk) | 0/223 | 0/223
Other Adverse Events (participants affected / at risk) | 0/223 | 0/223

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT02623335/Prot_SAP_000.pdf